CLINICAL TRIAL: NCT06214598
Title: Anti-Inflammatory Dietary Intervention in Breast Cancer Patients Receiving Aromatase Inhibitors
Brief Title: Anti-Inflammatory Diet in BRC Patients on Aromatase Inhibitors
Acronym: AID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Vesna Vucic, Principal Investigator, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AID5050
Record Dates: First submitted 2023-12-14; First posted 2024-01-19 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: AID project consists of a 3-arm clinical trial in BRC patients with 4-month nutritional intervention to assess the effects of personalized anti-inflammatory diet enriched with anti-inflammatory PUFA, or PUFA supplemental pills in 90 postmenopausal BRC patients receiving AI, randomly assigned in a ratio of 1:1:1 (diet:supplements:placebo). Since inflammation and oxidative stress are important promoters of cancer development and progression, we have chosen Fish oil and evening primrose oil as the richest sources of anti-inflammatory PUFA (n-3 and n-6). Anti-inflammatory diet enriched with PUFA and polyphenols was beneficial n many chronic diseases, and is named fatigue-reduction diet, especially relevant here as the fatigue is one of the most common side effects of AI. We will test the hypothesis that these interventions improve patients' nutritional status, QoL and clinical outcomes, by decreasing systemic inflammation and oxidative stress and reverting disrupted lipid metabolism.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo capusuls will be identical as supplement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AI Diet (Experimental): Personalised diet rich in whole grains high in fibres, vegetables (particularly leafy greens and tomatoes), polyphenol-rich fruits (berries), and n-3 FAs foods (fatty fish, nuts, seeds and oils)
  Interventions: Dietary Supplement: AI diet
- Supplements (Active Comparator): 2 gel capsules/d of fish oil (FO) + 3 gel capsules/d of evening primrose oil (EPO), containing 600 mg EPA, 400 mg DHA and 351 mg GLA + Standard diet: 55% carbohydrate, 15% protein and 30% fats
  Interventions: Dietary Supplement: Supplement
- Placebo (Placebo Comparator): Standard diet: 55% carbohydrate, 15% protein and 30% fats + placebo capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement — Supplements of anti-inflammatory oils rich in omega-3 and gamma-linolenic acid
  Arms: Supplements
Dietary Supplement: AI diet — diet rich in whole grains, healthy oils and polyphenols,
  Arms: AI Diet
Dietary Supplement: Placebo — Placebo caps with standard diet
  Arms: Placebo

SUMMARY:
This project aims to decrease undesirable side effects and increase qulaity of life of aromatase inhibitors therapy in breast cancer survivors, by anti-inflammatory diet or supplementation.

DETAILED DESCRIPTION:
With 2.1 million new breast cancer (BRC) cases each year globally, BRC is one of the biggest health challenges today. Available anticancer therapies have limited efficacy and are coupled with toxic side effects. Nutritional intervention can ameliorate undesirable effects, reduce exhaustion, psychological harm, and costs spent on treating these side effects. The proposed project AID aims to improve clinical outcome, quality of life (QoL) and survival rate in BRC patients on adjuvant endocrine therapy with aromatase inhibitors (AI) by nutritional interventions. In a three-arm randomised controlled nutritional trial involving 90 BRC patients who will receive either supplement or placebo pills (control group), or an anti-inflammatory diet for 4 months, along with the AI therapy, changes in nutritional status, QoL, biochemical and clinical parameters will be measured in comparison among three groups. The second goal is to establish cause-and-effect relationships among the clinical outcomes, nutritional status and biochemical parameters related to cancer, including inflammatory and redox status, plasma lipidome and polymorphism of fatty acid desaturase (FADS) genes. Introducing an effective nutritional intervention in BRC patients as an integral part of the multimodal therapeutic approach is the goal of this project.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45 to 70 years
* Postmenopausal women
* Histologically confirmed BRC, stage I to IIIa
* ER positive /HER2 negative
* Application of adjuvant hormone therapy with aromase inhibitors: 6 to 30 months
* Body mass index from 20 to 34.9 kg/m 2
* Able to understand the requirements of the study and provide written information consent

Exclusion Criteria:

* Metastatic or locally advanced disease
* HER2-positive tumors
* Presence of other malignant or serious chronic diseases
* Active infections
* Previous stroke or heart attack,
* Rheumatoid arthritis and other types of autoimmune diseases
* Presence of a significant neurological deficit
* Dementia
* Allergy to the ingredients of the dietary preparation or to fish, fish oil and nuts fruits.
* Allergies to evening primrose oil or other oils containing gamma-linolenic acid (borage, black currant)
* Use of lipid-lowering drugs (statins, Normolip)
* Current use of warfarin or other anticoagulants
* Corticosteroid therapy for the last month
* Use of dietary supplements based on fish oil, evening primrose, and flaxseed oils, omega 3-6-9 fatty acids, multivitamins with added omega-3 of fatty acids 3 months before the start of the study

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | baseline, 4 months, 1 year
  assessed through blood cells count
Nutritional status | baseline, 4 months, 1 year
  assessed through body mass index-BMI
Nutritional status | baseline, 4 months, 1 year
  assessed through body composition- lean tissue, fat tissue and body water (in kg)
Changes in Quality of life | baseline, 4 months
  assessed through the questionnaires FACT ES. The response scale is 5 point Likert-type scale (0- not at all, 4- very much).
Changes in Quality of life | baseline, 4 months
  assessed through the questionnaires EORTC QLQ-C30. All items are scored on a 4-point categorical scale ranging from 1- not at al to 4- very much, except the two items of the global quality of life which use a modified 7-point linear analogue scale ranging from 1- very bad to 7- excellent.
Changes in Quality of life | baseline, 4 months
  assessed through the questionnaires QLQ-BR23. All items are scored on a 4-point categorical scale ranging from 1- not at al to 4- very much.
Clinical outcome | baseline, 4 months, 1 year
  assessed through Laboratory analyses including BRC marker CA 15-3
Clinical outcome | baseline, 4 months, 1 year
  assessed through potential complications and side-effects

SECONDARY OUTCOMES:
Inflammatory status | baseline, 4 months,
  levels of inflammatory markers IL-6, IL-8, IL-10 and TNF-α
Redox status | baseline, 4 months,
  total antioxidant status (TAS), total advanced oxidation protein products (AOPP), total oxidant status (TOS), all in micromol/L
Redox status | baseline, 4 months,
  superoxide dismutase (SOD)
Redox status | baseline, 4 months,
  thiobarbituric acid reactive substances (TBARS)
leptin and adiponectin | baseline, 4 months
  plasma levels of leptin and adiponectin
Fatty acid status | baseline, 4 months
  Fatty acid mol% of plasma phospholipids
Lipidomic analysis | baseline, 4 months
  LC-MS lipids analysis
FADS1/FADS2 | baseline
  Polymorphism of FADS1/FADS2 genes to test if the patient is homozygote with major or minor alleles or heterozygote for rs174537, rs174576 and rs174602

CONTACTS AND LOCATIONS:
Locations (2):
- Serbia (2):
  - Clinical Hospital Center Bezanijska kosa, Belgrade
  - Center of Research Excellence in Nutrition and Metabolism, Institute for Medical Research, University of Belgrade, Belgrade

IPD SHARING:
Plan to Share IPD: No